CLINICAL TRIAL: NCT04386226
Title: An Assessment of the Glyconutrient Ambrotose™ on Immunity, Gut Health, and Safety in Men and Women: a Placebo-controlled, Randomized Clinical Trial
Brief Title: An Assessment of the Glyconutrient Ambrotose™ on Immunity, Gut Health, and Safety in Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Mannatech, Inc (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO-FY2018-488
Record Dates: First submitted 2020-05-05; First posted 2020-05-13 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: Ambrotose; Immunity; Gut Health

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Control
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 2 grams Ambrotose LIFE (Experimental): 2 grams daily for 8 weeks
  Interventions: Dietary Supplement: Ambrotose LIFE
- 4 grams Ambrotose LIFE (Experimental): 4 grams daily for 8 weeks
  Interventions: Dietary Supplement: Ambrotose LIFE
- 2 grams Advanced Ambrotose (Active Comparator): 2 grams daily for 8 weeks
  Interventions: Dietary Supplement: Advanced Ambrotose
- 4 grams Advanced Ambrotose (Active Comparator): 4 grams daily for 8 weeks
  Interventions: Dietary Supplement: Advanced Ambrotose
- Placebo (Placebo Comparator): 4 grams Maltodextrin daily for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ambrotose LIFE — Ambrotose LIFE contains aloe vera extract inner leaf gel, arabinogalactin, ghatti gum, glucosamine hydrogen chloride, gum tragacanth, vitamin A, beta carotene, wakame algae extract, rice starch, RiFiber (rice bran), and Modified Citrus Pectin with Sodium Alginate.
  Arms: 2 grams Ambrotose LIFE; 4 grams Ambrotose LIFE
Dietary Supplement: Advanced Ambrotose — Advanced Ambrotose contains aloe vera extract inner leaf gel, arabinogalactan, ghatti gum, glucosamine hydrogen chloride, gum tragacanth, vitamin A, beta carotene, wakame algae extract, and rice starch
  Arms: 2 grams Advanced Ambrotose; 4 grams Advanced Ambrotose
Other: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
This study evaluates the impact of two Ambrotose products on immunity, gut health, and associated measures in healthy men and women. Subjects are randomly assigned in double-blind manner to one of five conditions: 1) 2 grams Advanced Ambrotose, 2) 4 grams Advanced Ambrotose, 3) 2 grams Ambrotose LIFE, 4) 4 grams Ambrotose LIFE, or 5) placebo. Subjects ingested their assigned condition daily for eight weeks.

DETAILED DESCRIPTION:
The product Ambrotose, which contains a blend of glyconutrients, has been used by human subjects for several years. It has been shown to enhance immunity, improve cognitive performance, and enhance antioxidant capacity. To date, the treatment with Ambrotose has been very well tolerated, with adverse events limited to "mild" or "self-limiting" or absent altogether.

This study evaluates the impact of two Ambrotose products on immunity, gut health, and associated measures in healthy men and women. Subjects are randomly assigned in double-blind manner to one of five conditions: 1) 2 grams Advanced Ambrotose, 2) 4 grams Ambrotose Advanced, 3) 2 grams Ambrotose LIFE, 4) 4 grams Ambrotose LIFE, or 5) placebo. Subjects ingested their assigned condition daily for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* must be physically active by participating in structured exercise at least twice per week for 30 or more minutes per session;
* not be pregnant

Exclusion Criteria:

* diagnosed cardiovascular disease
* diagnosed metabolic disease
* diagnosed neurological disease
* using nutritional supplements or medications known to impact immunity or gut health

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
general well-being (Short Form-12) | at baseline
  A 12-item questionnaire was used to measure functional health and well-being from the subject's point of view during their intervention. Scores range from 0 to 100, with higher scores representing better self-reported health
general well-being (Short Form-12) | at 4 weeks
  A 12-item questionnaire was used to measure functional health and well-being from the subject's point of view during their intervention. Scores range from 0 to 100, with higher scores representing better self-reported health
general well-being (Short Form-12) | at 8 weeks
  A 12-item questionnaire was used to measure functional health and well-being from the subject's point of view during their intervention. Scores range from 0 to 100, with higher scores representing better self-reported health
Self-reported psychological general well-being index | at baseline
  The Self-reported psychological general well-being index was used to assess subject's perceived well-being during their intervention. The index goes from 0 (worst possible level of well-being) to 110 (maximum level of well being)
The Self-reported psychological general well-being index was used to assess subject's perceived well-being during their intervention. The index goes from 0 (worst possible level of well-being) to 110 (maximum level of well being) | at 4 weeks
  The Self-reported psychological general well-being index was used to assess subject's perceived well-being during their intervention. The index goes from 0 (worst possible level of well-being) to 110 (maximum level of well being)
The Self-reported psychological general well-being index was used to assess subject's perceived well-being during their intervention. The index goes from 0 (worst possible level of well-being) to 110 (maximum level of well being) | at 8 weeks
  The Self-reported psychological general well-being index was used to assess subject's perceived well-being during their intervention. The index goes from 0 (worst possible level of well-being) to 110 (maximum level of well being)
Self-reported assessment of fatigue & associated variables | at baseline
  A visual analog scale in which the subject was asked to make a mark on a 100-mm scale to indicate how he/she felt in regards to the variable in question during their intervention with 0 being "not at all" and 100 being "the most"
Self-reported assessment of fatigue & associated variables | at 4 weeks
  A visual analog scale in which the subject was asked to make a mark on a 100-mm scale to indicate how he/she felt in regards to the variable in question during their intervention with 0 being "not at all" and 100 being "the most"
Self-reported assessment of fatigue & associated variables | at 8 weeks
  A visual analog scale in which the subject was asked to make a mark on a 100-mm scale to indicate how he/she felt in regards to the variable in question during their intervention with 0 being "not at all" and 100 being "the most"
White blood cell numbers | at baseline
  We determined the white blood cell numbers for each subject during their intervention.
White blood cell numbers | at 4 weeks
  We determined the white blood cell numbers for each subject during their intervention.
White blood cell numbers | at 8 weeks
  We determined the white blood cell numbers for each subject during their intervention.
Interleukin-10 (IL-10) level following blood incubation | at baseline
  IL-10 was measured following blood incubation with Roswell Park Memorial Institute (RPMI) medium for 6 hrs
Interleukin-10 (IL-10) level following blood incubation | at 4 weeks
  IL-10 was measured following blood incubation with Roswell Park Memorial Institute (RPMI) medium for 6 hrs
Interleukin-10 (IL-10) level following blood incubation | at 8 weeks
  IL-10 was measured following blood incubation with Roswell Park Memorial Institute (RPMI) medium for 6 hrs
Interleukin-6 (IL-6) level following blood incubation | at baseline
  IL-6 was measured following blood incubation with RPMI medium for 6 hrs
Interleukin-6 (IL-6) level following blood incubation | at 4 weeks
  IL-6 was measured following blood incubation with RPMI medium for 6 hrs
Interleukin-6 (IL-6) level following blood incubation | at 8 weeks
  IL-6 was measured following blood incubation with RPMI medium for 6 hrs
Interleukin-1beta (IL-1beta) level following blood incubation | at baseline
  IL-1beta was measured following blood incubation with RPMI medium for 6 hrs
Interleukin-1beta (IL-1beta) level following blood incubation | at 4 weeks
  IL-1beta was measured following blood incubation with RPMI medium for 6 hrs
Interleukin-1beta (IL-1beta) level following blood incubation | at 8 weeks
  IL-1beta was measured following blood incubation with RPMI medium for 6 hrs
Tumor Necrosis Factor alpha (TNFalpha) level following blood incubation | at baseline
  TNFalpha was measured following blood incubation with RPMI medium for 6 hrs
Tumor Necrosis Factor alpha (TNFalpha) level following blood incubation | at 4 weeks
  TNFalpha was measured following blood incubation with RPMI medium for 6 hrs
Tumor Necrosis Factor alpha (TNFalpha) level following blood incubation | at 8 weeks
  TNFalpha was measured following blood incubation with RPMI medium for 6 hrs
IL-10 level following blood incubation with lipopolysaccharide (LPS) | at baseline
  IL-10 was measured following blood incubation with RPMI medium containing lipopolysaccharide (final concentration 250 ng/mL) for 6 hrs
IL-10 level following blood incubation with lipopolysaccharide (LPS) | at 4 weeks
  IL-10 was measured following blood incubation with RPMI medium containing lipopolysaccharide (final concentration 250 ng/mL) for 6 hrs
IL-10 level following blood incubation with lipopolysaccharide (LPS) | at 8 weeks
  IL-10 was measured following blood incubation with RPMI medium containing lipopolysaccharide (final concentration 250 ng/mL) for 6 hrs
IL-6 level following blood incubation with LPS | at baseline
  IL-6 was measured following blood incubation with RPMI medium containing lipopolysaccharide (final concentration 250 ng/mL) for 6 hrs
IL-6 level following blood incubation with LPS | at 4 weeks
  IL-6 was measured following blood incubation with RPMI medium containing lipopolysaccharide (final concentration 250 ng/mL) for 6 hrs
IL-6 level following blood incubation with LPS | at 8 weeks
  IL-6 was measured following blood incubation with RPMI medium containing lipopolysaccharide (final concentration 250 ng/mL) for 6 hrs
IL-1beta level following blood incubation with LPS | at baseline
  IL-1beta was measured following blood incubation with RPMI medium containing lipopolysaccharide (final concentration 250 ng/mL) for 6 hrs
IL-1beta level following blood incubation with LPS | at 4 weeks
  IL-1beta was measured following blood incubation with RPMI medium containing lipopolysaccharide (final concentration 250 ng/mL) for 6 hrs
IL-1beta level following blood incubation with LPS | at 8 weeks
  IL-1beta was measured following blood incubation with RPMI medium containing lipopolysaccharide (final concentration 250 ng/mL) for 6 hrs
TNFalpha level following blood incubation with LPS | at baseline
  TNFalpha was measured following blood incubation with RPMI medium containing lipopolysaccharide (final concentration 250 ng/mL) for 6 hrs
TNFalpha level following blood incubation with LPS | at 4 weeks
  TNFalpha was measured following blood incubation with RPMI medium containing lipopolysaccharide (final concentration 250 ng/mL) for 6 hrs
TNFalpha level following blood incubation with LPS | at 8 weeks
  TNFalpha was measured following blood incubation with RPMI medium containing lipopolysaccharide (final concentration 250 ng/mL) for 6 hrs
Serum Zonulin levels | at baseline
  Zonulin from blood serum during the intervention was measured using an ELISA
Serum Zonulin levels | at 4 weeks
  Zonulin from blood serum during the intervention was measured using an ELISA
Serum Zonulin levels | at 8 weeks
  Zonulin from blood serum during the intervention was measured using an ELISA

SECONDARY OUTCOMES:
Dietary Intake | at baseline
  Dietary intake of subjects for 5-days prior to testing days was entered into Food Processor Pro software and analyzed for analyzed for total calories, macro- and micro-nutrient composition
Dietary Intake | at 4 weeks
  Dietary intake of subjects for 5-days prior to testing days was entered into Food Processor Pro software and analyzed for analyzed for total calories, macro- and micro-nutrient composition
Dietary Intake | at 8 weeks
  Dietary intake of subjects for 5-days prior to testing days was entered into Food Processor Pro software and analyzed for analyzed for total calories, macro- and micro-nutrient composition

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No